CLINICAL TRIAL: NCT06566300
Title: Autologous Nanofat Grafting by Injection Versus With Microneedling in Post-burn and Traumatic Atrophic Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dalia Ibrahim Halwag, Principal investigator, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nanofat scar
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: To evaluate the efficiency autologous nanofat injection versus autologous nanofat delivered by microneedling in management of post burn atrophic and traumatic scars.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injection of autologous nanofat grafting (Experimental): Two separate scars with similar properties or splitting of one large post-burn atrophic scar. One (part of the) scar will be treated by injection of autologous nanofat grafting and the other (part of the) scar will be treated by microneedling with autologous nanofat graft.
  Interventions: Procedure: injection of autologous nanofat grafting
- microneedling with autologous nanofat graft (Experimental): Two separate scars with similar properties or splitting of one large post-burn atrophic scar. One (part of the) scar will be treated by injection of autologous nanofat grafting and the other (part of the) scar will be treated by microneedling with autologous nanofat graft.
  Interventions: Procedure: microneedling with autologus nanofat graft

INTERVENTIONS:
Procedure: injection of autologous nanofat grafting — Injection of nanfat graft
  Arms: injection of autologous nanofat grafting
Procedure: microneedling with autologus nanofat graft — delivery of nanofat graft with microneedling
  Arms: microneedling with autologous nanofat graft

SUMMARY:
This study aims to evaluate the efficiency autologous nanofat injection versus autologous nanofat delivered by microneedling in management of post burn atrophic and traumatic scars.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females between 18-60 years old. 2. Post-burn or traumatic atrophic scar > 6 months duration (16). 3. Patients not receiving any treatments for the scar within the past 3 months.

Exclusion Criteria:

* 1. Patients with contractures, hypertrophic and keloid scars. 2. Patients with history of bleeding disorders or coagulopathy, or on anticoagulant therpy.

  3. Diabetes and other systemic diseases that may be complicated by the procedure.

  4. Pregnant and lactating females. 5. BMI less than 18.5 6. Patients with scars at the donor site

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
change in the scar by by the patient and observer scar assessment scale (POSAS). | 6 months after the proceedure
  patient and observer scar assessment scale score will be uesd

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Upon request and as compatible by ethical considerations
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon request and as compatible by ethical considerations